CLINICAL TRIAL: NCT01361373
Title: Dopamine Treatment in Children With Cerebral Palsy With Dystonia- A Double Blind Controlled Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Hilla Ben Pazi, MD, Shaare Zedek Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: -L- Dopa-Cerebral Palsy
Record Dates: First submitted 2010-06-06; First posted 2011-05-26 (Estimated); Last update posted 2011-05-27 (Estimated); Status verified 2011-05

CONDITIONS: Dystonic Cerebral Palsy
MeSH Terms: interventions — Dihydroxyphenylalanine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- DOPAMINE (Active Comparator): Sinemet up to 10 mg/kg/day
  Interventions: Drug: L- DOPA
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: L- DOPA — Sinemet up to 10 mg/kg/ day increasing gradually for 2 weeks
  Arms: DOPAMINE
Drug: placebo — placebo for 2 weeks
  Arms: Placebo

SUMMARY:
Background:

Cerebral palsy (CP) is the main cause of childhood immobility and is defined as a non progressive injury to the developing central nervous system in children younger than 3 years, resulting in neurological and musculoskeletal abnormalities. The main pathophysiological causes are encephalopathy of prematurity (periventricular leukomalacia) hypoxic ischemic encephalopathy. Infections, infracts and migration defects are other less common causes of CP. The brain injury leads to functional motor impairment impacting on daily activities commonly manifests as a movement disorder: pyramidal, leading to spasticity and extra-pyramidal leading to dystonia and chorea. In most cases extensive brain injury causes a mixed movement disorder. Dystonia is defined as involuntary muscle contractions causing twisting and abnormal postures. While the neurological underpinnings of CP remain unknown, a link between low dopamine and increased acetylcholine release has recently been reported in dystonia. Dopamine is considered the first line of treatment in children with dystonia and CP followed by anticholiergic treatment with trihexphenidyl. The recommendation of dopaminergic treatment is based on need to rule out dopamine-responsive-dystonia, a rare genetic disorder, and on single case study reporting improvement in CP. A double blind study support or refute the use of dopamine treatment for dystonic CP was never reported. Working hypothesis and

Aims:

In children with CP due to a clear underlying pathology, dopamine treatment will not improve daily function. Methods: the investigators will perform a double blinded randomized controlled crossover study. 50 children ages 4-18 years with a clear pathophysiological cause for CP will be enrolled. Each child will receive dopamine and placebo treatment for 2 weeks with a 2 week washout interval. Participants will be randomized into 2 groups; one will receive placebo followed by dopamine and the other vice versa. The primary outcome measure, goal-attainment-scale, and secondary outcome functional measures (such as box and blocks, 9 hole pegs, pronation/ supination, finger sequencing) will be assessed at the beginning and end of each treatment as well as parent questionnaires regarding satisfaction and side effects.

Expected results:

No functional improvement with dopamine treatment compared to placebo.

Importance:

supplying sufficient data to support or refute the use of dopamine treatment for dystonic CP.

Probable implications to Medicine:

this may lead to a change in medical treatment guidelines for children with CP.

ELIGIBILITY:
Inclusion Criteria:

* clear pathophysiological cause for CP
* disabling dystonia in upper limbs

Exclusion Criteria:

* significant contractures
* psychiatric disorder

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-05 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
QUEST quality of upper extremity skills test score before and after treatment | 2 years
  The QUEST is a measure designed to evaluate movement patterns and hand function in children with cerebral palsy. It is administered within a play context. Items are related to quality of movement, not to chronological age. There are 36 items assessing dissociated movements, grasp, protective extension, and weight bearing.

SECONDARY OUTCOMES:
box and blocks, 9 hole pegs, pronation/ supination, finger sequencing | 2 years
  Difference between test scores before and after treatment. Namely:
  * of box transfered per minute time to complete the 9 hole pegs insertion.
  * pronation/ supination per 20 seconds time to complete 5 finger sequencing rounds

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Derived] Pozin I, Bdolah-Abram T, Ben-Pazi H. Levodopa does not improve function in individuals with dystonic cerebral palsy. J Child Neurol. 2014 Apr;29(4):534-7. doi: 10.1177/0883073812473645. Epub 2013 Jan 24. PMID 23349519